CLINICAL TRIAL: NCT01799291
Title: Decision Making and Mental Health: Cognitive De-Biasing and the Assessment of Pediatric Bipolar Disorder
Brief Title: Cognitive De-Biasing and the Assessment of Pediatric Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2KR401204-MMJ
Record Dates: First submitted 2013-02-24; First posted 2013-02-26 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2013-09

CONDITIONS: Decision Making; Bipolar Disorder
Keywords: Decision Making; Pediatric Bipolar Disorder; Assessment; Intervention
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment: Decision Making Tutorial (Other): A brief presentation on mood disorders (i.e., Control condition) combined with the intervention (i.e., Treatment condition): a 20-minute training on decision-making errors and cognitive de-biasing strategies.
  Interventions: Behavioral: Decision Making Tutorial
- Control (No Intervention): A brief presentation about mood disorders.

INTERVENTIONS:
Behavioral: Decision Making Tutorial — A web-based presentation focused on key "cognitive de-biasing" strategies, including helping clinician participants: consider alternative diagnoses (e.g., symptom checklists); decrease reliance on memory (e.g., mnemonics); and incorporate Bayesian reasoning (e.g., actuarial approaches).
  Arms: Treatment: Decision Making Tutorial

SUMMARY:
The primary aim is to test the efficacy of a new intervention to improve clinical judgment. The investigators focus on the assessment of pediatric bipolar disorder (PBD), a controversial diagnosis with frequent diagnostic errors, by educating mental health professionals in common cognitive pitfalls and training them in recommended de-biasing strategies. The investigators hypothesize that the Treatment group will show higher diagnostic accuracy than the Control condition: Participants receiving the cognitive de-biasing intervention will be less likely to commit faulty heuristics and race/ethnicity bias. Secondary aims include soliciting feedback about whether the skills were useful when diagnosing the vignettes, and whether skills and cases seem clinically realistic.

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) of 100 participants will test the efficacy of a new intervention to improve clinical judgment.

Eligible participants will be licensed or currently supervised by a licensed mental health professional and have experience working with pediatric populations.

Participants will be randomly assigned to either Treatment or Control conditions. All participants receive a 5 minute pre-recorded presentation about mood disorders, then read several case vignettes and respond to questions regarding judgments about probable diagnoses and next clinical actions.

Study administration is Web-based via a secure portal. After answering questions to confirm eligibility and provide informed consent, participants will complete a background questionnaire. The Web software, Qualtrics, will randomize participants to watch a brief presentation on mood disorders (i.e., Control condition) versus the same presentation on mood disorders combined with the intervention (i.e., Treatment condition). The intervention is a 20-minute training on decision-making errors and cognitive de-biasing strategies.

Next, all participants review four clinical vignettes. Using only four vignettes reduces participant burden and maximizes response rate. Qualtrics presents the case vignettes in random orders.

After completing the last vignette and corresponding questions, participants in the treatment condition rate their experience of the intervention. These questions address the secondary study aims: (a) how participants will use these new techniques in their clinical practice; and, (b) how the investigators can tailor the intervention to make it even more user-friendly and appealing to clinical audiences.

ELIGIBILITY:
Inclusion Criteria:

* Participants need to be: (a) licensed or currently supervised by a licensed mental health professional; and, (b) have experience treating child and adolescent patient populations for mental health issues.

Exclusion Criteria:

* Not meeting criterion (a) or (b) above.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | one time, immediately following Web-based presentation(s)
  Participants in treatment and control conditions report vignette characters' probable diagnoses after reading each vignette. These diagnoses were rated on a 3-point Likert scale of (1 = inaccurate diagnosis, 2 = somewhat accurate, and 3 = accurate diagnosis) using criteria established by the research team (which includes expert diagnosticians).

SECONDARY OUTCOMES:
Clinician attitudes toward intervention | one time, immediately after Web-based intervention
  Participants in the treatment group complete a brief questionnaire (4 items) about their attitudes toward the cognitive de-biasing intervention. This measure describes different aspects of the intervention (e.g., how helpful it was in making diagnostic decisions), and requires participants to make ratings on a 6-point scale: (1) strong agree; (2) agree; (3) somewhat agree; (4) somewhat disagree; (5) disagree; and, (6) strong disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa M Jenkins, M.A., Principal Investigator — University of North Carolina, Chapel Hill; Eric A Youngstrom, Ph.D., Study Chair — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States